CLINICAL TRIAL: NCT02944292
Title: Prospective, Interventional Multicentre Study on the Effect of Deepening of Sedation on Intra-abdominal Pressure
Brief Title: Effect of Sedation on Intra-abdominal Pressure
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tartu University Hospital (Other)
Responsible Party: Principal Investigator, Joel Starkopf, Professor of Anaesthesiology and Intensive Care, Tartu University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16062
Record Dates: First submitted 2016-10-14; First posted 2016-10-25 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Intra-abdominal Hypertension
Keywords: Intra-abdominal pressure; Intra-abdominal hypertension
MeSH Terms: conditions — Intra-Abdominal Hypertension | interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All enrolled patients (Experimental): Study population:
  Adult, mechanically ventilated patients with IAP between 12 and 20 mmHg in at least two consecutive measurements, spontaneous breathing activity of at least 6 breaths/minute, RASS score between 0 and -4, if no contraindications to propofol administration are present and no other immediate interventions to reduce IAP are planned
  Intervention: Deepening of sedation Deepening of sedation will be achieved with a bolus of propofol followed by continuous infusion for one hour.
  Interventions: Procedure: Deepening of sedation; Drug: Propofol

INTERVENTIONS:
Procedure: Deepening of sedation — Deepening of sedation will be achieved with a bolus and subsequent continuous infusion of propofol.
Drug: Propofol — Propofol will be dosed according to lean body weight (LBW) for bolus administration and according to total body weight (TBW) for continuous infusion.
  All patients will receive a bolus of propofol 1 mg/kg LBW as a rapid infusion during one minute. Measurements will be made one minute after the ending of bolus infusion. Continuous infusion of propofol at a rate of 3 mg/kg/h will be started immediately following completion of measurements, not later than 5 minutes after bolus administration. The propofol infusion rate is decreased in case of hemodynamic instability by 1 mg/kg/h and until a minimum of 1 mg/kg/h, if needed. Maximum total dose of infusion of 5 mg/kg/h will not be exceeded (bolus not considered).

SUMMARY:
The purpose of this study is to evaluate the effect of deepening of sedation on intra-abdominal pressure in mechanically ventilated adult patients with intra-abdominal hypertension.

DETAILED DESCRIPTION:
The importance of intra-abdominal pressure (IAP) in critically ill patients has been addressed increasingly. Several studies have shown that elevated mean IAP is associated with adverse ICU outcomes. The prevalence of intra-abdominal hypertension (IAH) among critically ill patients is as high as 50% if defined according to maximal IAP and half of it if defined according to mean IAP. Development of IAH during ICU period is an independent risk factor for death. Considering such significant impact on patients' outcome, international conference of experts has agreed and published recommendations for treatment of IAH and abdominal compartment syndrome. Among others, deepening of sedation is suggested as treatment option. The recommendation is based on expert opinion; there are no controlled clinical studies available to support this approach. Importantly, recent studies have shown that deep sedation itself may be associated with worse outcome to patients. Treggiari et al suggest that a strategy of light sedation affords benefits with regard to reduction of intensive care unit stay and duration of ventilation without negatively affecting subsequent patient mental health or patient safety. Others have shown reduced ICU mortality as well as reduced incidence of ventilator-associated pneumonia in conjunction with light sedation.

This is a prospective, interventional, multicentre study. There will be no control group.

Study subjects:

Adult, mechanically ventilated patients with IAP between 12 and 20 mmHg in at least two consecutive measurements, spontaneous breathing activity of at least 6 breaths/minute, RASS score between 0 and -4, if no contraindications to propofol administration are present and no other interventions to reduce IAP are planned.

Study intervention:

Sedation deepening will be achieved with a bolus of propofol 1 mg/kg followed by continuous infusion of propofol 3 mg/kg/h for one hour. Patients previously receiving propofol infusion will receive supplemental propofol per protocol up to a maximum infusion rate of 5 mg/kg/h.

Series of measurements of IAP will be performed before (once) and after (repeatedly) intervention (deepening of sedation).

Deepness of sedation will be assessed with RASS score.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Mechanical ventilation
* IAP between 12 and 20 mmHg in at least two consecutive measurements within 1-12 h
* Spontaneous breathing activity of at least 6 breaths/minute
* RASS score between 0 and -4
* Physician-led sedation (if sedated; as opposed to nurse-led protocol)

Exclusion Criteria:

* Contraindication for propofol administration
* Contraindication for IAP measurement in supine position with head-of-bed at 0°
* Other intervention for reduction of IAP planned
* Previous propofol infusion rate >4 mg/kg/h

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Intra-abdominal pressure | At 30 minutes after the start of deepening of sedation (propofol bolus)

SECONDARY OUTCOMES:
Intra-abdominal pressure | After sedative bolus; at 1) 15, 2) 30, 3) 60 minutes after starting the continuous infusion of propofol
Richmond Agitation-Sedation Scale | After sedative bolus; at 1) 15, 2) 30, 3) 60 minutes after starting the continuous infusion of propofol
Spontaneous and total respiratory rate | After sedative bolus; at 1) 15, 2) 30, 3) 60 minutes after starting the continuous infusion of propofol
Tidal volume | After sedative bolus; at 1) 15, 2) 30, 3) 60 minutes after starting the continuous infusion of propofol
PEEP, Ppeak, Pplat | After sedative bolus; at 1) 15, 2) 30, 3) 60 minutes after starting the continuous infusion of propofol
Total number of vasopressor and inotrope boluses | During the intervention
  From the beginning of the bolus injection of propofol until the end of the continuous infusion of propofol
Maximal increase in dose of noradrenaline | During the intervention
  From the beginning of the bolus injection of propofol until the end of the continuous infusion of propofol
Mean arterial pressure | After sedative bolus; at 1) 15, 2) 30, 3) 60 minutes after starting the continuous infusion of propofol
Abdominal perfusion pressure | After sedative bolus; at 1) 15, 2) 30, 3) 60 minutes after starting the continuous infusion of propofol

CONTACTS AND LOCATIONS:
Overall Officials: Joel Starkopf, MD PhD, Study Director — Tartu University Hospital; University of Tartu; Annika Reintam Blaser, MD PhD, Study Director — University of Tartu
Locations (1):
- Tartu University Hospital, Tartu, Tartu, Estonia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Malbrain ML, Chiumello D, Pelosi P, Wilmer A, Brienza N, Malcangi V, Bihari D, Innes R, Cohen J, Singer P, Japiassu A, Kurtop E, De Keulenaer BL, Daelemans R, Del Turco M, Cosimini P, Ranieri M, Jacquet L, Laterre PF, Gattinoni L. Prevalence of intra-abdominal hypertension in critically ill patients: a multicentre epidemiological study. Intensive Care Med. 2004 May;30(5):822-9. doi: 10.1007/s00134-004-2169-9. Epub 2004 Feb 3. PMID 14758472
- [Background] Malbrain ML, Chiumello D, Pelosi P, Bihari D, Innes R, Ranieri VM, Del Turco M, Wilmer A, Brienza N, Malcangi V, Cohen J, Japiassu A, De Keulenaer BL, Daelemans R, Jacquet L, Laterre PF, Frank G, de Souza P, Cesana B, Gattinoni L. Incidence and prognosis of intraabdominal hypertension in a mixed population of critically ill patients: a multiple-center epidemiological study. Crit Care Med. 2005 Feb;33(2):315-22. doi: 10.1097/01.ccm.0000153408.09806.1b. PMID 15699833
- [Background] Reintam A, Parm P, Kitus R, Kern H, Starkopf J. Primary and secondary intra-abdominal hypertension--different impact on ICU outcome. Intensive Care Med. 2008 Sep;34(9):1624-31. doi: 10.1007/s00134-008-1134-4. Epub 2008 May 1. PMID 18446319
- [Background] Cheatham ML, Malbrain ML, Kirkpatrick A, Sugrue M, Parr M, De Waele J, Balogh Z, Leppaniemi A, Olvera C, Ivatury R, D'Amours S, Wendon J, Hillman K, Wilmer A. Results from the International Conference of Experts on Intra-abdominal Hypertension and Abdominal Compartment Syndrome. II. Recommendations. Intensive Care Med. 2007 Jun;33(6):951-62. doi: 10.1007/s00134-007-0592-4. Epub 2007 Mar 22. PMID 17377769
- [Background] Treggiari MM, Romand JA, Yanez ND, Deem SA, Goldberg J, Hudson L, Heidegger CP, Weiss NS. Randomized trial of light versus deep sedation on mental health after critical illness. Crit Care Med. 2009 Sep;37(9):2527-34. doi: 10.1097/CCM.0b013e3181a5689f. PMID 19602975
- [Background] Rello J, Diaz E, Roque M, Valles J. Risk factors for developing pneumonia within 48 hours of intubation. Am J Respir Crit Care Med. 1999 Jun;159(6):1742-6. doi: 10.1164/ajrccm.159.6.9808030. PMID 10351912
- [Background] Malbrain ML, Cheatham ML, Kirkpatrick A, Sugrue M, Parr M, De Waele J, Balogh Z, Leppaniemi A, Olvera C, Ivatury R, D'Amours S, Wendon J, Hillman K, Johansson K, Kolkman K, Wilmer A. Results from the International Conference of Experts on Intra-abdominal Hypertension and Abdominal Compartment Syndrome. I. Definitions. Intensive Care Med. 2006 Nov;32(11):1722-32. doi: 10.1007/s00134-006-0349-5. Epub 2006 Sep 12. PMID 16967294
- Available data/document: Study Protocol — https://drive.google.com/open?id=0B-XpW352z4ZJMFdseHNwTWI2clU